CLINICAL TRIAL: NCT06268184
Title: Effect of Omega 3 Supplementation on Nutritional Status and Oxidative Stress in Children and Adolescents With End Stage Renal Disease on Regular Hemodialysis
Brief Title: Effect of Omega 3 on Oxidative Stress and Nutritional Status of Children on Regular Dialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, NohaSayed Ahmed Hamed Esmaeil, assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: omega3 in oxidative stress
Record Dates: First submitted 2024-01-29; First posted 2024-02-20 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Intervention Model Description: group 1: 30 children with ESRD receive omega 3 supplementation group 2:15 children with ESRD receive lpacebo
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- omega 3 (Active Comparator): D3LAB syrup each 5 ml contain :EPA 825 mg and DHA 550 mg each child receive 3.6 ml every day for 6 months
  Interventions: Dietary Supplement: D3 LAB SYRUP
- placebo (Placebo Comparator): Placebo capsules contain only the standard ingredients of soft gelatin capsules (gelatin, water, glycerin, and vitamin E in minute amounts as preservatives).
  Interventions: Dietary Supplement: placebo syrup

INTERVENTIONS:
Dietary Supplement: D3 LAB SYRUP — omega 3 suplementation
  Arms: omega 3
Dietary Supplement: placebo syrup — placebo syrup contains purified water, glycerin, xanthan gum, tween 80, methyl paraben, propyl paraben, sorbitol solution70% and apple flavor.
  Arms: placebo

SUMMARY:
evaluaion the effects of oral omega-3 supplementation on nutritional status and oxidative stress in pediatric patients with end stage renal disease on regular hemodialysis

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is a medically challenging and economically demanding health issue that adds to child morbidity and mortality.

The prevalence of pediatric CKD has been reported to be ranging from 15 to 74.7 cases per million children.

With an earlier age of onset of CKD, there is a greater risk of comorbidities associated with the disease including: malnutrition, growth.

retardation, joint pain, dental problems, hypertension, dyslipidemia and cardiovascular disease.

Kidney wasting disease is a common and serious complication of CKD, affects approximately one-third of end stage renal disease (ESRD) patients on hemodialysis. Contributing factors to this malnutrition include poor appetite, various co-morbidities, dietary restrictions, inflammation, infection, metabolic acidosis and oxidative stress. Oxidative stress (OS), defined as disturbances in the pro-

/antioxidant balance, is harmful to cells due to the excessive generation of highly reactive oxygen (ROS) and nitrogen (RNS) species.When the balance is not disturbed, OS has a role in physiological adaptations and signal transduction. The kidney is a highly metabolic organ, rich in oxidation reactions in mitochondria, which makes it vulnerable to damage caused by OS, in turn, OS is associated with kidney disease progression. Several complications of CKD are linked to increased levels of OS. Also, in ESRD, increased OS is associated with complications such as hypertension, atherosclerosis, inflammation, and anemia. The 'oxidative' link between CKD and its complications is achieved through several mechanisms, such as uremic toxin-induced endothelial nitric oxide synthase (eNOS) uncoupling and increased nicotinamide adenine dinucleotide phosphate-oxidases [NADPH oxidases (NOX)] activity. but also antioxidant losses due to dietary restrictions, diuretics use, protein energy wasting, and/or decreased intestinal absorption.

In CKD patients, lifestyle factors, such as aerobic exercise and dietary interventions, have been shown to exert anti-inflammatory effects. however, the adherence for CKD patients is often poor, thus leading to pharmacological therapy as a potential alternative. The use of statins, and angiotensin-converting enzyme inhibitors, as well as angiotensin II type 1 blockers, have been shown to exert some anti-inflammatory effects. In addition to the conventional therapy, the use of supplements has gathered interest in scientific research. Numerous studies have shown the possibility of using compounds with anti-inflammatory and antioxidant activities in the treatment of CKD.

Omega-3 fatty acids including Eicosapentaenoic acid and docosahexaenoic acid can modify abnormal lipid metabolism, decrease platelet aggregation, and improve endothelium function, blood pressure, heart rate, oxidative stress, and inflammation. Patients with ESRD have substantially lower blood levels of n-3 polyunsaturated fatty acids (n-3 PUFA) compared with the general population, probably due to lower dietary intake, inflammation, malabsorption, metabolic changes, and loss of n-3 PUFA during the dialysis process.

ELIGIBILITY:
Inclusion Criteria:

* ESRD children and adolescents on regular hemodialysis for at least 3 months
* Age ranging from 6 to18 years.

Exclusion Criteria:

* Systematic disease other than CKD eg SLE
* Severe active infection.
* Allergies to any of the ingredients in omega-3 product used in this study (e.g. fish oil, bovine gelatin).
* Omega-3 fatty acid or any other antioxidants consumption within the last 6 months.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
decrease oxidative stress | 6 months
  measured by assessment of serum level of Human Thiobarbituric Acid Reactive Substances (TBARS)
increase antioxidant activity | 6 months
  measured by assessment of serum level of Human Glutathione peroxidase (GSH-Px)
improvement of nutritional status assessed by anthropometric measurements. | 6 months
  including weight measure in kilograms ,height in meters, BMI calculated by division of weight on (height in meters)2
mid upper arm circumference in centimeters | 6 months
  improvement of nutritional status assessed by anthropometric measurements.
triceps skin fold thickness in millimeter's | 6 months
  improvement of nutritional status assessed by anthropometric measurements.
improvement of nutritional status assessed by Bioelectrical Inbody Analysis(BIA) | 6 months
  including fat mass index ( FMI)
improvement of nutritional status assessed by Bioelectrical Inbody Analysis(BIA) | 6 months
  fat free mass index (FFMI)
improvement of nutritional status assessed by Bioelectrical Inbody Analysis(BIA) | 6 months
  total body water percentage (TBW%)
improvement of nutritional status assessed by Bioelectrical Inbody Analysis(BIA) | 6 months
  Basal metaboic rate (BMR)
improvement of nutritional status assessed by Bioelectrical Inbody Analysis(BIA) | 6 months
  muscle mass percentage (MM%)
improvement of nutritional status assessed by laboratory investigations. | 6 months
  serum albumin level
s. ionized calcium level | 6 months
s.phosphorus level | 6 months
alkaline phosphatase level | 6 months
parathormone hormone level | 6 months
25(oh)vitamin D level | 6 months
  improvement of nutritional status assessed by laboratory investigations.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No